CLINICAL TRIAL: NCT05145062
Title: An Observational Long-term Safety and Efficacy Follow-up Study After Ex-vivo Gene Therapy With BIVV003 in Participants With Severe Sickle Cell Disease (SCD) or With ST-400 in Participants With Transfusion-dependent Beta-thalassemia (TDT) With Autologous Hematopoietic Stem Cell Transplant
Brief Title: Long - Term Follow Up of Sickle Cell Disease and Beta-thalassemia Subjects Previously Exposed to BIVV003 or ST-400.
Status: Active, not recruiting | Type: Observational
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: LTS16653
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Blood and Lymphatic Diseases
Keywords: Sickle Cell Disease (SCD), Beta-thalassemia (TDT)
MeSH Terms: conditions — Lymphatic Diseases; Anemia, Sickle Cell; beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BIVV003 Cohort: All participants treated in parent and future studies with BIVV003
  Interventions: Drug: BIVV003
- ST-400 Cohort: All participants treated in parent studies with ST-400
  Interventions: Drug: ST-400

INTERVENTIONS:
Drug: BIVV003 — Solution for intravenous administration
  Other Names: SAR445136
  Groups: BIVV003 Cohort
Drug: ST-400 — Solution for intravenous administration
  Groups: ST-400 Cohort

SUMMARY:
Primary Objectives:

Long-term safety of BIVV003 in participants with severe sickle cell disease (SCD) and ST- 400 in participants with transfusion-dependent beta-thalassemia (TDT)

Secondary Objectives:

* Long-term efficacy of the biological treatment effect of BIVV003 in SCD
* Long-term efficacy of the clinical treatment effect of BIVV003 on SCD-related clinical events
* Long-term efficacy of the biological treatment effect of ST-400 in TDT
* Long-term efficacy of the clinical treatment effect of ST-400 in TDT

DETAILED DESCRIPTION:
The total study duration is up to 15 years of follow-up post BIVV003 and/or ST-400 infusion.

ELIGIBILITY:
Inclusion Criteria:

* Received treatment with BIVV003 or ST-400 in one of the parent studies (ACT16222, ST- 400-01) or any future studies with BIVV003
* Capable of giving signed informed consent (and if applicable assent)

Exclusion Criteria:

* Unable to comply with study visit schedule or study procedures
* Any other reason that, in the opinion of the Investigator or Medical Monitor, would render the participant unsuitable for participation in the study The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All participants who received BIVV003 in one of the primary parent or future studies or ST-400 in the ST-400-01 parent study and agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2038-07-14 (Estimated); Study Completion 2038-07-14 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to 15 years
  Number of participants with serious adverse events and adverse events related to BIVV003 or ST-400, including new malignancy, new incidence or exacerbation of neurologic or rheumatologic or autoimmune or hematologic disorder, or new incidence of infection potentially related to BIVV003 or ST-400
Overall Survival | Up to 15 years
  Duration from first dose of study medication to death

SECONDARY OUTCOMES:
Change in hemoglobin levels | Up to 15 years
  Long-term change in levels of hemoglobin F, hemoglobin S and total hemoglobin (BIVV003 cohort), long term change in levels of hemoglobin F and total hemoglobin (ST-400 cohort)
Change in hemolysis markers | Up to 15 years
  Long-term change in markers of hemolysis, including reticulocyte count, lactate dehydrogenase, haptoglobin, and serum bilirubin, over time in the BIVV003 cohort
Frequency of severe vaso-occlusive crises | Up to 15 years
  Percentage of participants with severe vaso-occlusive crises, including acute pain crisis, acute chest syndrome, priapism, and splenic sequestration, in the BIVV003 cohort
Frequency and severity of SCD-related clinical events | Up to 15 years
  Percentage of participants with SCD-related clinical events (e.g., acute renal failure, acute stroke) in the BIVV003 cohort
Red blood cell transfusions | Up to 15 years
  Number and total volume of red blood transfusions in the BIVV003 and ST-400 cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics
Locations (7):
- United States (7):
  - UCSF Benioff Children's Hospital, Oakland, California
  - University of California Davis Health System, Sacramento, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No